CLINICAL TRIAL: NCT02229383
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Once Weekly Exenatide Therapy Added to Titrated Basal Insulin Glargine Compared to Placebo Added to Titrated Basal Insulin Glargine in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Basal Insulin Glargine With or Without Metformin
Brief Title: Phase III Study to Evaluate Safety and Efficacy of Added Exenatide Versus Placebo to Titrated Basal Insulin Glargine in Inadequately Controlled Patients With Type II Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5553C00002; 2014-003502-33 (EudraCT Number)
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Exenatide; Diabetes drug; Treatment efficacy; Placebo; Metabolism; Cardiovascilar metabolic
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Exenatide 2 mg 1 time per week + titrated basal insulin glargine with or without metformin
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Placebo 2 mg 1 time per week + titrated basal insulin glargine with or without metformin
  Interventions: Drug: Exenatide matching placebo

INTERVENTIONS:
Drug: Exenatide — 2 mg weekly suspension injection
  Arms: Exenatide
Drug: Exenatide matching placebo — Once weekly Placebo injection
  Arms: Placebo

SUMMARY:
Study D5553C00002 is a multicenter, randomized, double-blind, placebo-controlled, parallel group, Phase 3 study to compare the safety and efficacy of exenatide once weekly (EQW) added to titrated basal insulin glargine with or without metformin to placebo added to titrated basal insulin glargine with or without metformin in patients with type 2 diabetes mellitus (T2DM). Eligible patients will be randomized at Visit 5 (Day 1) to receive either EQW added to titrated basal insulin glargine, with or without metformin ≥1500 mg/day, or placebo added to titrated basal insulin glargine, with or without metformin ≥1500 mg/day, during the 28-week treatment period.

ELIGIBILITY:
Inclusion criteria:

* Has a diagnosis of Type 2 Diabetes Mellitus (T2DM)
* Has HbA1c of 7.5% to 12.0%, inclusive, at Visit 1 (Screening).
* Has fasting plasma glucose (FPG) concentration <280 mg/dL (15.6 mmol/L) at Visit 1 (Screening)
* Treated with basal insulin glargine at a dose of ≥20 units/day once daily for at least 6 weeks prior to Screening, in combination with diet and exercise alone or in combination with:

  1. a stable dose of metformin (≥1500 mg/day) for at least 8 weeks prior to Visit 1
  2. a stable dose of metformin (≥1500 mg/day) for at least 8 weeks prior to Visit 1 (Screening) and a stable dose of sulfonylurea for at least 8 weeks prior to the Screening visit

Exclusion criteria:

* Serum calcitonin concentration ≥40 pg/mL (≥40 ng/L) at Visit 1 (Screening)
* History of, or currently have, acute or chronic pancreatitis, or have triglyceride concentrations ≥500 mg/dL (≥5.65 mmol/L) at Visit 1
* Positive serological test for hepatitis B or hepatitis C

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2014-09-06 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2016-08-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (59):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Muscle Shoals, Alabama
  - Research Site, Tempe, Arizona
  - Research Site, Chino, California
  - Research Site, Chula Vista, California
  - Research Site, El Cajon, California
  - Research Site, Fresno, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Hills, California
  - Research Site, Tustin, California
  - Research Site, West Hills, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Brooksville, Florida
  - Research Site, Chiefland, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, North Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Franklin, Indiana
  - Research Site, Newton, Kansas
  - Research Site, Monroe, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Hazelwood, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Haddon Heights, New Jersey
  - Research Site, Mooresville, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greer, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Dakota Dunes, South Dakota
  - Research Site, Johnson City, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Clinton, Utah
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Manassas, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Port Orchard, Washington
- Hungary (13):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gödöllő
  - Research Site, Gyula
  - Research Site, Komárom
  - Research Site, Létavértes
  - Research Site, Pécs
  - Research Site, Sátoraljaújhely
  - Research Site, Szeged
  - Research Site, Szekszárd
- Poland (7):
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Oświęcim
  - Research Site, Poznan
  - Research Site, Torun
  - Research Site, Zamość
  - Research Site, Zgierz
- Romania (7):
  - Research Site, Baia Mare
  - Research Site, Bucharest
  - Research Site, Galati
  - Research Site, Oradea
  - Research Site, Ploieşti
  - Research Site, Tg Mures
  - Research Site, Timișoara
- Slovakia (9):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Štúrovo
- South Africa (7):
  - Research Site, Bloemfontein
  - Research Site, Kempton Park
  - Research Site, Krugersdorp
  - Research Site, Paarl
  - Research Site, Pretoria
  - Research Site, Somerset West
  - Research Site, Worcester

REFERENCES:
- [Derived] Guja C, Frias JP, Suchower L, Hardy E, Marr G, Sjostrom CD, Jabbour SA. Safety and Efficacy of Exenatide Once Weekly in Participants with Type 2 Diabetes and Stage 2/3 Chronic Kidney Disease. Diabetes Ther. 2020 Jul;11(7):1467-1480. doi: 10.1007/s13300-020-00815-z. Epub 2020 Apr 18. PMID 32306296
- [Derived] Guja C, Frias JP, Somogyi A, Jabbour S, Wang H, Hardy E, Rosenstock J. Effect of exenatide QW or placebo, both added to titrated insulin glargine, in uncontrolled type 2 diabetes: The DURATION-7 randomized study. Diabetes Obes Metab. 2018 Jul;20(7):1602-1614. doi: 10.1111/dom.13266. Epub 2018 Mar 25. PMID 29473704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 107 centers globally between 06 September 2014 and 29 August 2016.
Pre-assignment Details: The study had a Screening Visit, an 8-week insulin dose optimization phase, followed by a 28-week randomized, double-blind treatment phase. A total of 464 participants were randomized and entered the double-blind Treatment Period. Of which, 3 participants from 1 center in the United States have been excluded from analyses.
Groups:
- Exenatide: Exenatide 2 milligram (mg) 1 time per week + titrated basal insulin glargine with or without metformin.
- Placebo: Placebo (matching with exenatide) 1 time per week + titrated basal insulin glargine with or without metformin.
Period: Overall Study
Arm/Group | Exenatide | Placebo
Started | 232 | 229
Received Treatment | 231 | 229
Safety Analysis Set | 231 | 229
Intent-to-treat (ITT) Analysis Set | 230 | 228
Completed | 212 | 207
Not Completed | 20 | 22
Not completed — Adverse Event | 7 | 4
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Did not receive treatment | 1 | 0
Not completed — Other | 3 | 8

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants is comprised of the ITT analysis set: All randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline hemoglobin A1c (HbA1c) assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Placebo | Total
Number analyzed (Participants) | 230 | 228 | 458
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (9.04) | 57.5 (10.28) | 57.7 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 122 | 239
  Male | 113 | 106 | 219
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Black Or African American | 19 | 28 | 47
  Native Hawaiian Or Other Pacific Islander | 1 | 0 | 1
  Other | 1 | 4 | 5
  White | 204 | 194 | 398

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 28
Description: To compare the change from baseline in HbA1c achieved with exenatide once weekly (EQW) added to titrated basal insulin glargine to placebo added to titrated basal insulin glargine, with or without metformin, after 28 weeks of double-blind treatment. SU= sulfonylurea.
Time Frame: Baseline to Week 28
Population: The ITT analysis set included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline HbA1c assessment. Only participants with data available for analysis are presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of HbA1c
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 230 | 228
Percentage of HbA1c | -0.96 [-1.12 to -0.81] | -0.22 [-0.38 to -0.07]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Treatment, region, baseline HbA1c (< or ≥ 9.0%), baseline SU-use, week, treatment by week interaction as fixed factors; baseline value as covariate; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-0.94 to -0.54], Standard Error of Mean 0.101

2. Secondary Outcome: Change in Body Weight From Baseline to Week 28
Description: To compare the change from baseline in body weight achieved with EQW added to titrated basal insulin glargine to placebo added to titrated basal insulin glargine, with or without metformin, after 28 weeks of double-blind treatment.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 230 | 228
kilogram | -1.04 [-1.54 to -0.53] | 0.48 [-0.02 to 0.98]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.52, 95% CI 2-sided [-2.19 to -0.85], Standard Error of Mean 0.341

3. Secondary Outcome: Change From Baseline to Week 28 in 2-hour Postprandial Glucose After a Standard Meal Tolerance Test (MTT)
Description: To compare the change from baseline in 2-hour postprandial glucose after a standard MTT achieved with EQW added to titrated basal insulin glargine to placebo added to titrated basal insulin glargine, with or without metformin, after 28 weeks of double-blind treatment.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: milligram per deciliter
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 230 | 228
milligram per deciliter | -28.73 [-40.0 to -17.45] | -0.96 [-12.41 to 10.48]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment, region, baseline HbA1c (< or ≥ 9.0%), baseline SU-use (yes vs. no) as fixed factors; baseline value as covariate; Mean Difference (Final Values) = -27.76, 95% CI 2-sided [-39.07 to -16.45], Standard Error of Mean 5.754

4. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0% at Week 28
Description: To compare the percentage of participants achieving HbA1c <7.0% between EQW added to titrated basal insulin glargine to placebo added to titrated basal insulin glargine, with or without metformin, after 28 weeks of double-blind treatment.
Time Frame: Baseline to Week 28
Population: The ITT analysis set included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline HbA1c assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 230 | 228
Percentage of participants | 32.6 [26.6 to 38.7] | 7.0 [3.7 to 10.3]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline HbA1c (<9.0% or ≥9.0%) and baseline SU-use (yes vs. no); Difference in percentages = 25.6

5. Secondary Outcome: Change From Baseline to Week 28 in Daily Insulin Dose
Description: To compare the change from baseline in daily insulin dose achieved with EQW added to titrated basal insulin glargine to placebo added to titrated basal insulin glargine, with or without metformin, after 28 weeks of double-blind treatment.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 230 | 228
Units | 1.6 [0.1 to 3.1] | 3.5 [2.0 to 5.1]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p = 0.074, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-4.1 to 0.2], Standard Error of Mean 1.08

6. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0% at Week 28, No Weight Gain at Week 28, and No Major Hypoglycemia Over 28 Weeks
Description: To compare the percentage of participants achieving HbA1c <7.0% at Week 28, no weight gain at Week 28, and no major hypoglycemia over 28 weeks between EQW added to titrated basal insulin glargine to placebo added to titrated basal insulin glargine, with or without metformin.
Time Frame: Baseline to Week 28
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 230 | 228
Percentage of participants | 22.2 [16.8 to 27.5] | 2.2 [0.3 to 4.1]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline HbA1c (<9.0% or ≥9.0%) and baseline SU-use (yes vs. no); Difference in percentages = 20.0

7. Secondary Outcome: Change in Seated Systolic Blood Pressure From Baseline to Week 28
Description: To compare the change from baseline in seated systolic blood pressure achieved with EQW added to titrated basal insulin glargine to placebo added to titrated basal insulin glargine, with or without metformin, after 28 weeks of double-blind treatment.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter of mercury
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 230 | 228
millimeter of mercury | -2.5 [-4.4 to -0.7] | -0.7 [-2.6 to 1.1]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p = 0.110, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-4.0 to 0.4], Standard Error of Mean 1.13

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) up to Week 28
Description: Safety analysis set included all participants who received at least 1 dose of randomized study medication. All-Cause Mortality is reported for the overall study period, including the off-treatment period; Serious and Other adverse event data is reported for the on-treatment period.
Arm/Group | Exenatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/231 | 1/229
Serious Adverse Events (participants affected / at risk) | 11/231 | 11/229
Other Adverse Events (participants affected / at risk) | 40/231 | 36/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=231) | Placebo (N=229)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=231) | Placebo (N=229)
Nausea (Gastrointestinal disorders) | 12 (13) | 9 (10)
Injection site nodule (General disorders) | 12 (14) | 1 (1)
Urinary tract infection (Infections and infestations) | 18 (25) | 15 (21)
Blood creatine phosphokinase increased (Investigations) | 5 (6) | 13 (15)

LIMITATIONS AND CAVEATS:
Please note that the data from 4 subjects enrolled at one site were omitted due to potential scientific misconduct at that site. Study conclusions remain unchanged.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 30 days prior to submission for publication or presentation, Authors shall provide Sponsor with such material for its review. Sponsor shall have 30 days to comment. If requested by Sponsor, Authors shall withhold material for an additional 90 days to allow for the taking of measures to establish its proprietary rights. No publication or presentation shall be made unless and until any information determined at Sponsor's sole discretion to be Confidential has been removed.